CLINICAL TRIAL: NCT03623048
Title: Effect of Propolis and Pomegranate Extract Mouthwash on Taste Alteration, Salivary pH and Antibacterial Activity in High Caries Risk Patients
Brief Title: Effect of Natural Antibacterial Mouthwash on Taste, Salivary pH and Bacteria in High Caries Risk pt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Randa Abdelrahman, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-08-04
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Decay, Dental
MeSH Terms: conditions — Dental Caries | interventions — Chlorhexidine; hexitol; Sodium Chloride; Saline Solution; Propolis; pomegranate fruit rind

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Propolis extract (Experimental): intervention
  Interventions: Other: Propolis extract
- Pomegranate extract (Experimental): intervention
  Interventions: Other: pomegranate extract
- Chlorhexidine (Active Comparator): comparator
  Interventions: Other: chlorhexidine
- Saline (Placebo Comparator): comparator
  Interventions: Other: saline

INTERVENTIONS:
Other: chlorhexidine — antibacterial and anti-inflammatory mouthwash
  Other Names: hexitol
  Arms: Chlorhexidine
Other: saline — anti-inflammatory cleansing mouthwash
  Other Names: NaCl solution
  Arms: Saline
Other: Propolis extract — antibacterial mouthwash
  Arms: Propolis extract
Other: pomegranate extract — antibacterial mouthwash
  Arms: Pomegranate extract

SUMMARY:
Evaluate the effect of propolis extract mouthwash and pomegranate extract mouthwash on taste alteration, salivary pH and antibacterial activity against streptococcus mutans in high caries risk patients.

DETAILED DESCRIPTION:
This study will be carried out to evaluate and compare the effect of propolis extract mouthwash and pomegranate (botanical name: Punica granatum) extract mouthwash on taste alteration, salivary pH and antibacterial activity against streptococcus mutans in high caries risk patients.

Thats by taking unstimulated saliva samples at the morning before using the mouthwash, then taking another one after using the mouthwash and finally after 7 days, to make a bacterial culture and measure the salivary pH by a digital pH meter and evaluate taste changes by a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* High caries risk patients defined according to American Dental Association (ADA)
* Systematically healthy
* Not taking any medication interfering with saliva secretion
* Subjects who signed informed consent
* Age range from 17-50 years

Exclusion Criteria:

* Subjects suffering from any medical or systematic disease
* Smokers
* Pregnant females
* Allergy to any of the mouthwash ingredients
* Patients older than 50 years

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Taste alteration | One week
  taste changes will be measured by a questionnaire

SECONDARY OUTCOMES:
Salivary pH | one week
  salivary pH will be measured by digital pH meter